CLINICAL TRIAL: NCT07072988
Title: A Multicenter, Prospective, Observational, Open-label Study to Evaluate the Benefit of Corticoid Sparing in Elderly With Generalized AntiRAch Myasthenia Gravis Treated With IV or SC Efgartigimod
Brief Title: Evaluate the Benefit of Corticoid Sparing in Elderly With Generalized AntiRAch Myasthenia Gravis Treated With IV or SC Efgartigimod
Acronym: OPTIMAGE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-PP-08
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly with Generalized Anti-AChR Myasthenia Gravis Treated with IV or SC Efgartigimod (Experimental)
  Interventions: Drug: Efgartigimod

INTERVENTIONS:
Drug: Efgartigimod — Administration of efgartigimod, a neonatal Fc receptor (FcRn) antagonist, given either intravenously (IV) or subcutaneously (SC) to treat patients with generalized Anti-AChR Myasthenia Gravis.

SUMMARY:
Generalized Myasthenia Gravis (gMG) is a rare chronic autoimmune disorder causing muscle weakness and fatigue, primarily due to autoantibodies that disrupt neuromuscular junction function. The most common antibodies target nicotinic acetylcholine receptors (AChR), with others such as anti-MuSK and anti-LRP4 being less prevalent. The conventional gMG treatments include acetylcholinesterase inhibitors, corticosteroids, immunosuppressant and, in case of myasthenic crisis, plasma exchange (PLEX) and intravenous immunoglobulins (IVIG). Treatment aims to achieve minimal manifestation status (MMS), but many patients face persistent symptoms or side effects. Corticosteroids, while effective, carry significant risks, especially for long-term use, such as, increased infection and cardiovascular risks, chronic conditions like hypertension, diabetes, and osteoporosis and quality of life impacts, including weight gain and mood changes. Elderly patients, who form the majority of the gMG population, are particularly vulnerable due to age-related comorbidities, which limit treatment options and prolong corticosteroid reliance. This contributes to increased mortality, disability, and dependency. Efgartigimod (EFG), a novel therapeutic targeting the neonatal Fc receptor (FcRn), accelerates degradation of pathogenic IgG antibodies, including anti-AChR. Clinical trials demonstrated its efficacy and safety in reducing antibody levels, improving muscle strength, and enhancing quality of life. Both intravenous (IV) and subcutaneous (SC) forms are effective and well tolerated. Approved in the United States and subsequently in Japan and Europe, EFG became available in France in 2023. The present multicenter observational study aims to evaluate the real-life impact of EFG in elderly gMG patients struggling with corticosteroid side effects or comorbidity exacerbations. The objectives of this study include the assessing EFG's ability to enable corticosteroid reduction and monitoring improvements in gMG symptoms, quality of life, comorbidities, and overall health.

This approach highlights a shift towards targeted therapies that balance efficacy with reduced treatment-related burdens for vulnerable gMG populations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥65 years
* Diagnosed with gMG with confirmed documentation and supported by a physical exam and confirmed seropositivity for AChR-Abs.
* Meets the clinical criteria as defined by the Myasthenia Gravis Foundation of America (MFGA) for generalized MG class IIa, Iib, IIIa, IIIb.
* Patient suitable for efgartigimod treatment
* MG-ADL score ≥ 2
* Treated with high (>50mg/daily) or intermediate (20-50mg/daily) dose of oral corticosteroids (prednisone or prednisolone) and in stable dose of concomitant treatments for at least three months (changes of anticholinesterase therapy are permitted).
* Patient that has developed at least one of the following iatrogenic comorbidities after the introduction of intermediate or high dose of oral corticosteroids: type 2 diabetes; arterial hypertension; overweight; sleep disorders; irritability and/or Patient experiencing a documented worsening of at least one of the following comorbidities after the introduction of intermediate or high dose of corticosteroids, including type 2 diabetes; arterial hypertension; overweight; sleep disorders; irritability
* Capable of understanding the written informed consent, and providing signed, dated, and witnessed written informed consent
* Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures
* Patient affiliated to a European social security system

Exclusion Criteria:

* Any current mental condition (psychiatric disorder, senility, or dementia) that, in the opinion of the investigator, may affect study compliance or prevent understanding of the aims, investigational procedures, or possible consequences of the study; and/or patient with a Mini-mental State Examination (MMSE) <28.
* History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Ongoing malignancy including solid tumors, hematologic malignancies and in situ carcinoma (except basal cell and squamous cell carcinomas of the skin, or in situ carcinoma of the cervix uteri that have been completely excised and cured)
* Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening
* Vaccination with live or live-attenuated vaccines within the 6 weeks
* Patient already treated with anti-complement (wash-out period 3 months) or anti-FcRN (wash-out period 3 months), anti-CD20 (wash-out period 6 months) and PLEX (wash-out period 1 month)
* Patient with end-stage disease or with a disease that will enable him to be evaluated and/or treated
* Patient protected by law, under guardianship or curator ship, or not able to participate in a clinical study according to the article L.1121-16 of the French Public Health Code.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
evaluate at 12 months the change from baseline in the mean dose of corticosteroids in gMG patients switched to EFG | 12 mois
  evaluate at 12 months the change from baseline in the mean dose of corticosteroids in gMG patients switched to EFG

SECONDARY OUTCOMES:
change in percentage of patients in low dose of corticosteroid (<20mg) at 12 months | 12 months
  change from baseline of the percentage of patient treated with <20 mg of corticosteroids
change in percentage of patients in intermediate dose of corticosteroid (≥20 mg - ≤50 mg) at 12 months | 12 months
  change from baseline of the percentage of patient treated with ≥20 mg - ≤50 mg of corticosteroids
change in percentage of patients in high dose of corticosteroid (≥ 50mg) at 12 months | 12 months
  change from baseline of the percentage of patient treated with >50 mg of corticosteroids
change in Glucocorticoid Toxicity Index (GTI) at 12 months | 12 months
  change from baseline in GTI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France